CLINICAL TRIAL: NCT02090530
Title: Precision Cancer Medicine for Advanced Cancer Through High-throughput Sequencing
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sameek Roychowdhury, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-13053; NCI-2014-00632 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-03-07; First posted 2014-03-18 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: Cancer Genomics; Tumor Sequencing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Biopsy Whole Blood Serum Buccal Smear Plasma Formalin Fixed Paraffin Embedded (FFPE) Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Cancer Patients: Individuals with advanced or refractory cancer must be identified by study personnel or their treating physician, deemed eligible for this study, and voluntarily agree to be enrolled in this protocol through an informed consent. Biospecimen collection includes a fresh tumor biopsy, previously obtained tumor specimens or blocks (if available), whole blood, serum, plasma and buccal smear.
  Interventions: Other: Biospecimen collection

INTERVENTIONS:
Other: Biospecimen collection — Specimens to be collected include a fresh tumor biopsy, previously obtained tumor specimens or blocks (if available), whole blood, serum, plasma and buccal smear.

SUMMARY:
Precision Cancer Medicine for Advanced Cancer Through High-throughput Sequencing

DETAILED DESCRIPTION:
This study supports the collection of tumor specimens for CLIA-certified genomic testing and research testing in parallel. CLIA-certified tests have established measurements of accuracy and precision which allow for return of results. This study does not involve treatment, only testing, which could be used to meet eligibility criteria in other trials or therapies. This study includes a registry for longitudinal evaluation of patients whose cancer has FGFR mutations such as cholangiocarcinoma, pancreatic cancer, and others (telehealth).

ELIGIBILITY:
Inclusion Criteria:

1. A histologically or cytologically confirmed diagnosis of cancer
2. Patients with any malignancy.
3. Patients must have tumor suitable for research tumor biopsy (as assessed by trained specialists in interventional radiology) and Patients are medically fit to undergo a tissue biopsy or surgical procedure to get tumor tissue OR If Patients do not have a tumor suitable for biopsy but have another tissue available for molecular evaluation.

   OR Patients are undergoing standard of care surgeries or procedures where fresh specimens will be first used for routine pathologic assessment and only then will leftover tissue be used for research purposes.
4. Procedure-specific signed informed consent prior to initiation of any study-related procedures.
5. Women and minorities are included in this protocol.
6. Patients with multiple malignancies remain eligible.
7. Patients with an inherited cancer syndrome or a medical history suggestive of an inherited cancer syndrome remain eligible.

Exclusion Criteria:

1. It is the enrolling study physicians discretion to decide if a patient is not fit enough to undergo tissue biopsy.
2. Patients who are incarcerated are not eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or refractory cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-11-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants receiving new therapy based on study findings | Up to 24 Months
  Impact on clinical care

SECONDARY OUTCOMES:
Average number of days to return results | Up to 24 months
  Determine average number of days for return of results

CONTACTS AND LOCATIONS:
Overall Officials: Sameek Roychowdhury, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krook MA, Bonneville R, Chen HZ, Reeser JW, Wing MR, Martin DM, Smith AM, Dao T, Samorodnitsky E, Paruchuri A, Miya J, Baker KR, Yu L, Timmers C, Dittmar K, Freud AG, Allenby P, Roychowdhury S. Tumor heterogeneity and acquired drug resistance in FGFR2-fusion-positive cholangiocarcinoma through rapid research autopsy. Cold Spring Harb Mol Case Stud. 2019 Aug 1;5(4):a004002. doi: 10.1101/mcs.a004002. Print 2019 Aug. PMID 31371345
- See also: The Jamesline — http://cancer.osu.edu